CLINICAL TRIAL: NCT03764696
Title: The Effect of Maternal Long Term High Flow Oxygen Administration During Labor on Umbilical Cord Blood Gases
Brief Title: Maternal Oxygen Administration for Fetal Distress II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yunhai Chuai, Clinical Professor of Obstetrics and Gynecology, Principal Investigator, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYH002
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Oxygen Inhalation Therapy; Labour; Fetal Distress
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- air, the first and second stage of labor (No Intervention): Patients randomized to the group will receive room air.
  The therapy will continue until after delivery
- oxygen, the first and second stage of labor (Experimental): Patients randomized to the group will receive oxygen administered by high flow facemask oxygen at 10 L/min oxygen.
  The therapy will continue until after delivery
  Interventions: Device: tight-fitting simple facemask

INTERVENTIONS:
Device: tight-fitting simple facemask — Oxygen will be administered by facemask at 10 L/min oxygen. The therapy will continue until after delivery
  Arms: oxygen, the first and second stage of labor

SUMMARY:
Supplementary oxygen is routinely administered to patients, even those with adequate oxygen saturations, in the belief that it increases oxygen delivery. However, oxygen delivery depends not just on arterial oxygen content but also on perfusion.

Maternal oxygen administration has been used in an attempt to lessen fetal distress by increasing the available oxygen from the mother. However, the effect of supplemental maternal oxygen therapy on fetal acid base status has been debated for more than seven decades.

The investigators found the use of 2 L/min maternal oxygen during the second stage of labor did not adversely affect either the umbilical artery pH value or the fetal heart rate (FHR) pattern distribution.

ELIGIBILITY:
Inclusion Criteria:

at term (>37 weeks, <42 weeks), singleton, cephalic presentation, spontaneous or induced labor, normal labor, category I FHR tracings, 2 to 3 cm of cervical dilation in nulliparity, 1 to 2 cm of cervical dilation in multipara, informed consent.

Exclusion Criteria:

respiratory or cardiovascular disease, diabetes mellitus or insulin-treated gestational diabetes mellitus, hypertension or preeclampsia, oligohydramnios, fetal growth restriction, placental abruption, cephalopelvic disproportion, meconium-stained amniotic fluid, tachysystole, having received O2, uterine incision (myomectomy or perforation), anemia, fever, chorioamnionitis, tobacco or alcohol use, disorders in oxygen saturations, hypotension, uncomfortable with facemask.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cord arterial pH values | within 30 to 60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), blood gas sample will be obtained.
Cord arterial partial pressure of oxygen | within 30 to 60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), blood gas sample will be obtained.
Cord arterial partial pressure of carbon dioxide | within 30 to 60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), blood gas sample will be obtained.
Cord venous pH values | within 30 to 60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), blood gas sample will be obtained.
Cord venous partial pressure of oxygen | within 30 to 60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), blood gas sample will be obtained.
Cord venous partial pressure of carbon dioxide | within 30 to 60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), blood gas sample will be obtained.

SECONDARY OUTCOMES:
Rate of abnormal fetal heart tracing | at 1 minute after birth

OTHER OUTCOMES:
Rate of cesarean delivery | at 1 minute after birth
Rate of assisted vaginal delivery | at 1 minute after birth
Apgar score less than 7 | at 1 and 5 minutes after birth
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from 0 to 2, then summing up the five values thus obtained. The resulting Apgar score ranges from 0 to 10. The five criteria are summarized using words chosen (Appearance, Pulse, Grimace, Activity, Respiration). The infant is given a score of 0, 1 or 2. The scores are added up and the total sum is their Apgar score.
  The test is generally done at one and five minutes after birth, and may be repeated later if the score is and remains low. Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low.
Rate of serious neonatal morbidity or death | within 28 days of birth
Cord arterial plasma liquid chromatography mass spectrometry analysis | within 30 to 60 seconds of birth
  The systematic identification and quantitation of all the metabolic products (mainly endogenous small molecule compounds with relative molecular weight within 1000 Da) of cord arterial plasma under oxygen and room air conditions. Immediately after delivery (within 30-60 seconds of birth), blood plasma sample will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Yunhai Chuai, Dr, Principal Investigator — Sixth Medical Center, Chinese PLA General Hospital; Fang Chuai, Principal Investigator — Sixth Medical Center, Chinese PLA General Hospital
Locations (3):
- China (3):
  - Department of Obstetrics and Gynecology, PLA Strategic Support Force Characteristic Medical Center, Beijing
  - Department of Obstetrics and Gynecology, Seventh Medical Center, Chinese PLA General Hospital, Beijing
  - Department of Obstetrics and Gynecology, Sixth Medical Center, Chinese PLA General Hospital, Beijing

REFERENCES:
- [Background] Chuai F, Dong T, Liu Y, Jiang W, Zhang L, Chen L, Chuai Y, Zhou Y. The effect of intrapartum prolonged oxygen exposure on fetal metabolic status: secondary analysis from a randomized controlled trial. Front Endocrinol (Lausanne). 2023 Jun 27;14:1204956. doi: 10.3389/fendo.2023.1204956. eCollection 2023. PMID 37441500
- [Background] Chuai Y, Jiang W, Zhang L, Chuai F, Sun X, Peng K, Gao J, Dong T, Chen L, Yao Y. Effect of long-duration oxygen vs room air during labor on umbilical cord venous partial pressure of oxygen: a randomized controlled trial. Am J Obstet Gynecol. 2022 Oct;227(4):629.e1-629.e16. doi: 10.1016/j.ajog.2022.05.028. Epub 2022 May 14. PMID 35580635